CLINICAL TRIAL: NCT01507246
Title: A Pain Relief Trial Utilizing the Infiltration of a Multivesicular Liposome Formulation Of Bupivacaine, EXPAREL®: A Phase 4 Health Economic Trial in Adult Patients Undergoing Open Colectomy
Brief Title: Adult Patients Undergoing Open Colectomy MA402S23B303
Acronym: IMPROVE-Open
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Collaborators: Registrat-Mapi (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: MA402S23B303
Record Dates: First submitted 2011-10-23; First posted 2012-01-10 (Estimated); Results first posted 2013-05-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Bowel Obstruction
Keywords: open colectomy
MeSH Terms: conditions — Intestinal Obstruction | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV morphine sulfate (Active Comparator): Standard of Care (SOC), dosage variable, administered intravenously via PCA pump postsurgically, as need.
  Interventions: Drug: IV morphine sulfate
- EXPAREL (bupivacaine liposome injectable suspension) (Experimental): EXPAREL(R), dosage 266 mg, diluted with 0.9% saline to a total volume of 40 cc.
  Interventions: Drug: EXPAREL (bupivacaine liposome injectable suspension)

INTERVENTIONS:
Drug: IV morphine sulfate — Patients in this group will receive IV morphine sulfate via PCA pump, as needed. The PCA pump will be set up postsurgically as soon as possible and prior to the patient leaving the PACU or immediately upon transfer to the floor if the stay in the PACU is less than one hour.
  Other Names: morphine sulfate (or Sponsor-approved equivalent)
  Arms: IV morphine sulfate
Drug: EXPAREL (bupivacaine liposome injectable suspension) — Patients in this group will receive 266 mg EXPAREL diluted with preservative free 0.9% normal saline to a total volume of 30 cc and administered via wound infiltration prior to wound closure. When not contraindicated, 30 mg IV ketorolac will be given at the end of surgery. If not indicated, an IV non-steroidal anti-inflammatory drug (NSAID) may be substituted per the site's standard of care.
  All patients will be offered rescue analgesia, as needed.
  Other Names: bupivacaine free base
  Arms: EXPAREL (bupivacaine liposome injectable suspension)

SUMMARY:
This study is designed to compare the standard of care against EXPAREL(R) to determine if total opioid consumption is reduced when using EXPAREL, therefore possibly reducing total hospitalization costs.

DETAILED DESCRIPTION:
This is a phase 4, prospective, sequential, open-label study designed to evaluate the efficacy, safety, and health economic benefits of intraoperative local wound infiltration with EXPAREL compared with postsurgical administration of standardized intravenous (IV) morphine sulfate or sponsor-approved equivalent for postsurgical analgesia in adult patients undergoing open colectomy with general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age and older.
* Patients scheduled to undergo open segmental colectomy with planned primary anastamosis, as defined by cecectomy, right hemicolectomy, resection of transverse colon, left hemicolectomy, or sigmoidectomy.
* Ability to provide informed consent, adhere to study visit schedule, and complete all assessments.

Exclusion Criteria:

* Patients with a history of hypersensitivity or idiosyncratic reactions or intolerance to any local anesthetic, opioid, or propofol.
* Patients who abuse alcohol or other drug substance.
* Patients with severe hepatic impairment.
* Patients currently pregnant or who may become pregnant during the course of the study.
* Patients with any psychiatric, psychological, or other condition that the Investigator feels may make the patient an inappropriate candidate for this clinical study.
* Patients who have participated in an EXPAREL study within the last 30 days.
* Patients who have received an investigational drug within 30 days prior to study drug administration, or planned administration of another investigational product or procedure during the patient's participation in this study.
* Patients who undergo any concurrent surgical procedure during the ileostomy reversal surgery

In addition, the patient will be ineligible if he/she meets the following criteria during surgery:

* Patients who have any concurrent surgical procedure.
* Patients with unplanned multiple segmental resections or large intestine.
* Patients who have unplanned, temporary or permanent colostomies, ileostomies, or the like placed.
* Patients who receive intraoperative administration of opioids (other than fentanyl or analogs) or an other analgesic, local anesthetics, or anti-inflammatory agents.
* Patients who receive Entereg(R).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cohen, M.D., Principal Investigator — Atlanta Colon and Rectal Surgery
Locations (1):
- Atlanta Colon and Rectal Surgery, Riverdale, Georgia, United States

REFERENCES:
- [Derived] Cohen SM, Vogel JD, Marcet JE, Candiotti KA. Liposome bupivacaine for improvement in economic outcomes and opioid burden in GI surgery: IMPROVE Study pooled analysis. J Pain Res. 2014 Jun 24;7:359-66. doi: 10.2147/JPR.S63764. eCollection 2014. PMID 25018650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment Dec 13, 2011 to July 3, 2012
Pre-assignment Details: open-label, sequential study with two treatment groups. Patients were to be excluded if they met certain intraoperative exclusion criteria.
Groups:
- PCA/Opioid Group: Group receiving standardized IV morphine sulfate or Sponsor-approved equivalent via PCA pump postsurgically, as needed.
- EXPAREL Group: Group receiving EXPAREL
Period: Overall Study
Arm/Group | PCA/Opioid Group | EXPAREL Group
Started | 20 | 22
Completed | 18 | 21
Not Completed | 2 | 1
Not completed — Required different surgical procedures | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCA/Opioid Group | EXPAREL Group | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 32
  >=65 years | 5 | 5 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 54.1 (15.77) | 52.6 (17.51) | 53.3 (16.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Burden
Description: Total opioid consumed (IV and PO) postsurgically until the hospital discharge order is written or through Day 30, whichever is sooner.
Time Frame: Wound closure to time hospital discharge order written or Day 30, whichever is sooner
Population: Per protocol
Measure: Mean (Standard Deviation); unit: mg
Groups:
- PCA/Opioid Group: Group receiving standardized IV morphine or Sponsor-approved equivalent via PCA pump postsurgically, as need.
- EXPAREL: Group receiving EXPAREL
Arm/Group | PCA/Opioid Group | EXPAREL
Number analyzed (Participants) | 18 | 21
mg | 115.00 (113.27) | 56.76 (74.04)
Statistical Analysis 1: Comparison: PCA/Opioid Group vs EXPAREL; Null hypothesis: Mean ratio of geometric least-squares mean for each group is identical; Test type: Superiority or Other; p = 0.0251, least-squares mean ratio; Ratio of geometric means = 2.62, 95% CI 2-sided [1.14 to 6.03] — Group 1 represents the numerator

2. Primary Outcome: Health Economic Benefits - Total Cost of Hospitalization
Description: Total cost of hospitalization until the time hospital discharge order is written or through Day 30, whichever is sooner.
Time Frame: Wound closure to time hospital discharge order written or Day 30, whichever is sooner.
Population: per protocol
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | PCA/Opioid Group | EXPAREL
Number analyzed (Participants) | 18 | 21
dollars | 11850.28 (6600.90) | 8766.07 (1048.95)
Statistical Analysis 1: Comparison: PCA/Opioid Group vs EXPAREL; Null hypothesis = distribution of costs is identical between the two groups; Test type: Superiority or Other; p = 0.02767, least-squares mean ratio; Ratio of geometric means = 1.24, 95% CI 2-sided [1.03 to 1.49] — Group 1 represents the numerator

3. Secondary Outcome: Incidence of Predefined Opioid-related Adverse Events
Description: The incidence of predefined opioid-related adverse events
Time Frame: From the time the informed consent is signed to the time hospital discharge order is written or through Day 30 (after surgery), which ever is sooner
Population: Per protocol.
Measure: Number; unit: Number of patients
Groups:
- PCA/Opioid Group: Group receiving standardized IV morphine or Sponsor-approved equivalent via PCA pump postsurgically, as needed.
Arm/Group | PCA/Opioid Group | EXPAREL
Number analyzed (Participants) | 18 | 21
Number of patients | 0 | 0

4. Primary Outcome: Health Economic Benefits - Length of Stay
Description: Length of stay (LOS), recorded in hours and converted to days with one decimal of precision, defined as the time of completion of the wound closure until the hospital discharge order is written or through Day 30, whichever is sooner.
Time Frame: Up to Day 30
Population: All subjects analyzed, no censored events
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PCA/Opioid Group | EXPAREL Group
Number analyzed (Participants) | 18 | 21
days | 4.9 [3.9 to 6.7] | 2.0 [1.9 to 3.0]

ADVERSE EVENTS:
Arm/Group | PCA/Opioid Group | EXPAREL Group
Serious Adverse Events (participants affected / at risk) | 4/18 | 5/21
Other Adverse Events (participants affected / at risk) | 4/18 | 7/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCA/Opioid Group (N=18) | EXPAREL Group (N=21)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Wound evisceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Drug Seeking Behavior (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCA/Opioid Group (N=18) | EXPAREL Group (N=21)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Post Procedural Hematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound Evisceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Creatine Increased (Investigations) | 1 (1) | 0 (0)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Therapy Regimen Changed (Surgical and medical procedures) | 1 (1) | 0 (0)
Wound Drainage (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No